CLINICAL TRIAL: NCT03087617
Title: Personalized Smoking Cessation Tool Based on Patient Lung CT Image
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imbio (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); University of Michigan (Other); Mayo Clinic (Other); HealthPartners Institute (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: R44CA203050 (NIH); R44CA203050 (NIH)
Record Dates: First submitted 2017-03-02; First posted 2017-03-22 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: University of Minnesota Office of Measurements Services will administer follow up calls to assess outcomes. Callers will be blinded to the arm to which the patients were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Usual Care (Active Comparator): Usual Care includes a lung cancer screening CT exam. Following the screen, a radiologist will analyze the CT scan image and send the results to the patient's Primary Care Physician (PCP). If the scan is read as a category 1 or 2 in the Lung Reporting and Data System (Lung-RADS), patients are provided a letter in the mail with their results. If the scan is read as a category 3, 4A, 4B, or 4X in Lung-RADS the patient will be contacted by their primary care physician's office and told to schedule a follow up appointment. Either in the letter or at the follow up appointment, patients will be given a Quitline number created specifically for this trial and maintained for the duration.
  Interventions: Other: Usual Care
- Usual Care + Imbio Smoking Cessation Report (Experimental): In this arm, patients will receive the Usual Care described above and will additionally be provided with the Report. In this arm, the Report will provide the Quitline number.
  Interventions: Device: Imbio Smoking Cessation Report; Other: Usual Care
- Usual Care + Counseling (Active Comparator): In addition to the Usual Care described above, patients in this arm will participate in a 45 minute smoking cessation counseling session. Approximately three Tobacco Treatment Specialists will be trained to ensure consistent counseling methodology. Counselors will utilize a patient centered approach grounded in Motivational Interviewing skills to elicit perceived benefits for stopping smoking and to enhance self-efficacy for stopping. A major emphasis of a call is to enroll the caller in formal cessation programs and/or convince them to use FDA approved medication as part of a quit attempt. Study participants who desire further smoking cessation support after their session will be connected with the appropriate organization.
  Interventions: Behavioral: Smoking Cessation Counseling; Other: Usual Care
- Usual Care + Imbio Smoking Cessation Report + Counseling (Experimental): In addition to the Usual Care and Counseling described above, patients in this arm will also receive the Report.
  Interventions: Device: Imbio Smoking Cessation Report; Behavioral: Smoking Cessation Counseling; Other: Usual Care

INTERVENTIONS:
Device: Imbio Smoking Cessation Report — Research coordinators at the University of Michigan and HealthPartners will be provided access to the research version of LDA via an Imbio website. Following consent and lung screen, research coordinators will manually upload the study participants' images and download a resulting Report. Radiologists have been designated at both sites to review and approve the Report prior to mailing to participants. The Report will include information including the percent of damaged lung volume.
  Other Names: Smoking Cessation Report; Report
  Arms: Usual Care + Imbio Smoking Cessation Report; Usual Care + Imbio Smoking Cessation Report + Counseling
Behavioral: Smoking Cessation Counseling — 45 minute counseling session with a tobacco treatment specialist.
  Arms: Usual Care + Counseling; Usual Care + Imbio Smoking Cessation Report + Counseling
Other: Usual Care — Usual Care for Lung Cancer Screening patients.

SUMMARY:
Imbio is developing a Smoking Cessation Report (Report) that includes data analysis from a CT lung cancer screening exam. This randomized controlled (RCT) trial will clinically validate the Report's effectiveness at motivating smokers to call a Quitline.

DETAILED DESCRIPTION:
Imbio is developing a Smoking Cessation Report (Report) that includes data analysis from a CT lung cancer screening exam. This randomized controlled (RCT) trial will clinically validate the Report's impact on: (a) Lung screening participants' motivation to make a quit attempt by calling a Quitline, and (b) the effectiveness of a 45-minute telephone smoking cessation counseling session for motivating an actual quit attempt and abstinence. The RCT will enroll approximately 400 randomly selected participants from lung screening programs at HealthPartners and University of Michigan. Participants will be randomly assigned to one of four conditions: 1) Usual Care + quitline phone number (created specifically for the trial and maintained for the length of the trial); 2) Usual Care + Report (Report will list Quitline number) 3) Usual Care + Counseling, or 4) Usual Care + Report + Counseling. Follow up assessment calls will be conducted with participants at three weeks, three months, and six months following the mailing of the report.

ELIGIBILITY:
Inclusion Criteria:

* 30-pack year smoking history
* currently smoke OR quit within the last 15 years and a category 1 or 2 Lung-RADS scan

Exclusion Criteria:

* current use of smoking cessation medications
* scan read as a category 3, 4A, 4B or 4X in Lung-RADS
* unstable medical or psychiatric conditions
* current alcohol or drug use disorder
* past-month suicidal ideation
* past-year suicide attempt

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Health Partners, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Usual Care + Imbio Smoking Cessation Report | Usual Care + Counseling | Usual Care + Imbio Smoking Cessation Report + Counseling
Started | 79 | 80 | 82 | 80
Completed | 47 | 50 | 52 | 41
Not Completed | 32 | 30 | 30 | 39
Not completed — Lost to Follow-up | 32 | 30 | 30 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Usual Care + Imbio Smoking Cessation Report | Usual Care + Counseling | Usual Care + Imbio Smoking Cessation Report + Counseling | Total
Number analyzed (Participants) | 79 | 80 | 82 | 80 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (6) | 65 (6) | 65 (5.45) | 65 (6) | 65 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 52 | 38 | 166
  Male | 41 | 42 | 30 | 42 | 155
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 79 | 80 | 82 | 80 | 321

OUTCOME MEASURES:

1. Primary Outcome: Report's Impact on Calling a Quitline Number
Description: This outcome will be measured by whether the participant calls the Quitline number provided to them.
  ***Given logistical complexities, it was never the intention to measure this outcome on a participant level, but rather to compare the arms as different groups to see if there is a difference in the number of calls received for each groups Quitline number, which was automatically monitored. Unfortunately, it because apparent that the monitored Quitline numbers were subject to many robocalls and that data because too unreliable to be analyzed.
Time Frame: 3 weeks after intervention.
Population: Given logistical complexities, it was never the intention to measure this outcome on a participant level, but rather to compare the arms as different groups to see if there is a difference in the number of calls received for each groups Quitline number, which was automatically monitored. Unfortunately, it because apparent that the monitored Quitline numbers were subject to many robocalls and that data because too unreliable to be analyzed.
Arm/Group | Usual Care | Usual Care + Imbio Smoking Cessation Report | Usual Care + Counseling | Usual Care + Imbio Smoking Cessation Report + Counseling
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Report's Impact Making a Quit Attempt Measured Via Follow-up Phone Call
Description: This outcome will be measured by the participants' motivation to make a quit attempt and abstain from smoking. The question asked was: How ready are you to quit smoking?
  Answer options include:
  1. Not at all ready
  2. Slightly ready
  3. Moderately ready
  4. Very ready
Time Frame: 3 weeks after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Usual Care + Imbio Smoking Cessation Report | Usual Care + Counseling | Usual Care + Imbio Smoking Cessation Report + Counseling
Number analyzed (Participants) | 66 | 72 | 75 | 69
score on a scale | 2.73 (0.84) | 3.15 (0.90) | 2.92 (0.87) | 2.97 (0.92)

3. Primary Outcome: Report's Impact on Calling a Quitline Number
Description: This outcome will be measured by whether the participant calls the Quitline number provided to them.
Time Frame: 3 months after intervention
Population: ***Given logistical complexities, it was never the intention to measure this outcome on a participant level, but rather to compare the arms as different groups to see if there is a difference in the number of calls received for each groups Quitline number, which was automatically monitored. Unfortunately, it because apparent that the monitored Quitline numbers were subject to many robocalls and that data because too unreliable to be analyzed.
Arm/Group | Usual Care | Usual Care + Imbio Smoking Cessation Report | Usual Care + Counseling | Usual Care + Imbio Smoking Cessation Report + Counseling
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Report's Impact on Calling a Quitline Number
Description: This outcome will be measured by whether the participant calls the Quitline number provided to them.
Time Frame: 6 months after intervention
Population: as for outcome 3
Arm/Group | Usual Care | Usual Care + Imbio Smoking Cessation Report | Usual Care + Counseling | Usual Care + Imbio Smoking Cessation Report + Counseling
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Report's Impact Making a Quit Attempt Measured Via Follow-up Phone Call
Description: as for outcome 2
Time Frame: 3 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Usual Care + Imbio Smoking Cessation Report | Usual Care + Counseling | Usual Care + Imbio Smoking Cessation Report + Counseling
Number analyzed (Participants) | 53 | 53 | 54 | 46
score on a scale | 2.75 (0.92) | 3.08 (0.92) | 2.61 (0.98) | 3.07 (0.90)

6. Primary Outcome: Report's Impact Making a Quit Attempt Measured Via Follow-up Phone Call
Description: as for outcome 2
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Usual Care + Imbio Smoking Cessation Report | Usual Care + Counseling | Usual Care + Imbio Smoking Cessation Report + Counseling
Number analyzed (Participants) | 47 | 50 | 52 | 41
score on a scale | 2.85 (0.88) | 3.00 (0.93) | 2.80 (0.93) | 3.07 (0.96)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care | Usual Care + Imbio Smoking Cessation Report | Usual Care + Counseling | Usual Care + Imbio Smoking Cessation Report + Counseling
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/80 | 0/82 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/80 | 0/82 | 0/80
Other Adverse Events (participants affected / at risk) | 0/79 | 0/80 | 0/82 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03087617/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03087617/ICF_001.pdf